CLINICAL TRIAL: NCT00602134
Title: A Pharmacokinetic Study to Assess the Single-Dose Bioequivalence of a Potential Generic Formulation of a 6-Mercaptopurine 50 mg Tablet Compared to a Marketed 6-Mercaptopurine 50 mg Tablet, Purinethol®, When Administered to Healthy Male Subjects, in the Fasted State
Brief Title: Bioequivalence Study of 6-Mercaptopurine Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Director, Drug Regulatory Affairs and Medical Affairs, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 439-09
Record Dates: First submitted 2007-09-19; First posted 2008-01-28 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Mercaptopurine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 6-Mercaptopurine

SUMMARY:
The objective of this study was to assess the bioequivalence of a potential generic 6-mercaptopurine 50 mg tablet formulation compared with GlaxoSmithKline Purinethol® (mercaptopurine) 50-mg scored tablets following a single 50 mg oral dose administered in the fasted state.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on physical examination, medical history, or clinical laboratory results.
* Must voluntarily consent.

Exclusion Criteria:

* Must not have a known history of thiopurine methyltransferase deficiency or family history.
* Must not have a history of elevated uric acid or gout.
* Must not be currently using allopurinol.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2002-11; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | Baseline, two period, 3 day washout

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Allison, MD, Principal Investigator — MDS Pharma Services
Locations (1):
- MDS Pharma Services, Phoenix, Arizona, United States